CLINICAL TRIAL: NCT05823844
Title: Improvement of Restorative Sleep and Post-surgical Insomnia Following Suvorexant Administration
Brief Title: Efficacy of Suvorexant on Post-operative Sleep Disturbance
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Paul Garcia, Associate Professor of Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAU4343
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Insomnia; Postoperative Delirium
Keywords: Sleep Disturbance; Insomnia; Sleep quality; Suvorexant
MeSH Terms: conditions — Emergence Delirium; Parasomnias; Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: This study is a parallel-group, double-blind, randomized trial where 92 subjects will to randomized 1:1 to either receive 20 mg Suvorexant or placebo (two tablets) and treatment as usual.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Raters and subjects will be blinded to treatment. At the study's completion (the last subject completes) the blind will be broken, and data will be turned over for analysis. A study physician will be available on call 24 hours to monitor patient safety issues that may arise during the hospitalization and they will have access to the blind. Furthermore, the Research Pharmacy will maintain the blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Suvorexant administration (Experimental): Subjects will receive 20 mg Suvorexant beginning the first in-hospital night ("day 0") and continuing for their hospital stay. If the dose is not well tolerated (e.g., daytime sleepiness), then the dose may be decreased to 10 mg of Suvorexant. For blinding purposes, each arm will receive two tablets (two 10 mg tablets or one 10 mg tablet and a placebo). Suvorexant will be administered beginning on the night after surgery and through the hospitalization period (it is estimated that stays will be 1-3 days; subjects will be followed for a maximum of 5 days).
  Interventions: Drug: Suvorexant
- Placebo administration (Placebo Comparator): Subjects will receive a placebo (two tablets) and treatment as usual. The placebo will be administered beginning on the night after surgery and through the hospitalization period (it is estimated that stays will be 1-3 days; subjects will be followed for a maximum of 5 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant — Suvorexant (Belsomra™) is an orexin receptor antagonist that will be administered as 2 tablets (10mg each) for a starting dose of 20mg. If the dose is not well tolerated (e.g., daytime sleepiness), then the dose may be decreased to 10 mg of Suvorexant.
  Other Names: Belsomra
  Arms: Suvorexant administration
Drug: Placebo — The placebo pill will look identical to Suvorexant and will be taken as 2 tablets.
  Arms: Placebo administration

SUMMARY:
The study is a parallel group, double blind, randomized trial. Subjects will be recruited from individuals undergoing elective surgery for orthopedic, abdominal, urologic, gynecologic or spine reasons. Out of 92 subjects, one experimental group of 46 subjects will receive 20 mg Suvorexant beginning the first in-hospital night ("day 0") and continuing for their hospital stay. If the dose is not well tolerated (e.g., daytime sleepiness), then the dose may be decreased to 10 mg of Suvorexant.

For blinding purposes each arm will receive two tablets (two 10 mg tablets or one 10 mg tablet and a placebo). The other control group of 46 subjects will receive placebo (two tablets) and treatment as usual.

DETAILED DESCRIPTION:
It is rare to get a good night's sleep in the hospital. Even routine patient care, including alarm systems, and too much light can lead to sleep disturbance. Failure to achieve enough high-quality sleep has been associated with decreased brain and heart function. The investigators aim to restore usual sleep patterns in hospitalized patients to have a positive influence on patient outcomes and healthcare costs. Suvorexant, the tested drug in our protocol, works on a different brain chemical system than most other sleep drugs, which may account for its ability to restore natural sleep. Suvorexant has been shown to reduce wakefulness during sleep by a reduction in long wake bouts. This reduction has a positive effect on sleep quality. In keeping with Suvorexant's established ability to decrease insomnia in outpatient settings, the investigators will assess its efficacy to improve sleep quality in the hospital environment in patients having surgery who have sleep disturbance. Suvorexant will be administered beginning on the night after surgery and through the hospitalization (it is estimated that stays will be 1-3 days; the investigators will set a maximum of 4 days). If the dose is not well tolerated (e.g., daytime sleepiness), then the dose may be decreased to 10 mg of Suvorexant. The investigators aim to study the participant's sleep patterns by using a self-wearable electroencephalography (EEG) recording device, the Sleep Profiler, and see patterns such as total sleep time or the stages of sleep such as rapid eye movement (REM), non-REM, etc. Additionally, the investigators hope to determine if concentration, attention, and general cognitive performance are improved as a result of better sleep. Promoting "natural sleep" may improve surgical recovery through the lessening of fatigue and improvements in brain health.

ELIGIBILITY:
Inclusion criteria:

* Aged 50 years to 90 years old.
* Patients getting elective surgeries for orthopedic reasons (e.g., hip or knee replacement), abdominal surgery (e.g., hernia repair, renal cancer), urologic or gynecologic surgery, and spine surgery with a projected inpatient stay of 24 hours or longer.
* Patients experiencing insomnia characterized by difficulties with sleep onset, early morning awakening, and/or sleep maintenance three or more times weekly over a three-month period for eligibility.

Exclusion criteria:

* Patients who undergo surgery and then are admitted to intensive care.
* Coronary artery bypass graft (CABG) or other cardiac surgeries.
* Intra-cranial surgery.
* Patients taking more than 60 mg of oxycodone or it's equivalent as outpatient
* Circadian rhythm disorders.
* High score in the Geriatric Depression Scale (GDS)
* Moderate to severe dementia (failed t-MoCa)
* Severe obstructive sleep apnea (OSA) (Apnea-hypopnea index (AHI)>30 and/or screen high risk)
* Patients receiving Cytochrome P-450 (CYP3) inhibitors or inducers (Inhibitors: clarithromycin, erythromycin, diltiazem, itraconazole, ketoconazole, ritonavir, verapamil, goldenseal, and grapefruit. Inducers: phenobarbital, phenytoin, rifampicin, St. John's Wort, and glucocorticoids).
* Vulnerable populations (i.e., children, pregnant women).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Total sleep time on day 0 (TST) | Day 0 of in-hospital stay after surgery
  Analysis will be adjusted for group baseline differences, including pre-existing cognitive impairment, medical co-morbidities, and the type and duration of surgery.

SECONDARY OUTCOMES:
Longitudinal trend of TST | Up to Day 5 post-surgery
  The longitudinal trend of TST over the five days will be measured using mixed-effect regression. Group, time (day 0-4), and group x time will be included as the fixed effects and a random intercept of subjects to account for within-subject correlation due to repeated measurement. Regression quotients will be reported.
Rate of attrition | Up to Day 5 post-surgery
  The rate of attrition over the 5 days will be measured. If any specific patterns are identified, inverse propensity treatment weighting will be performed to adjust the effect of nonrandom dropout.
Richards Campbell Self-Report Sleep Scale | Up to Day 5 post-surgery
  The Richards Campbell self-report sleep scale will be used to determine the quality of sleep each morning. This five-item, visual analogue scale was designed as an outcome measure for assessing the perception of sleep. The scale evaluates perceptions of depth of sleep, sleep onset latency, number of awakenings, time spent awake, and overall sleep quality. For each item, respondents are given a visual analogue scale and are asked to place a mark on the line indicating where their own experiences fit between two extremes (for example, the degree to which they received a "good night's sleep" or "a bad night's sleep"). Scale lines extend from 0 to 100 mm, and scores are calculated by measuring where responses fall on each line. A total score is obtained by summing each score out of 100 and dividing the total by five. Lower scores indicate a poorer quality of sleep (worse outcome).
Incidence of Delirium | Up to Day 5 post-surgery
  The 3-minute diagnostic interview for Confusion Assessment Method (CAM)-defined delirium (3D-CAM) is a brief verbal assessment tool that can be used to test for delirium. For all items, if the subject's answer is 'incorrect', 'yes', 'don't know', 'no response', or 'non-sensical response', then the appropriate (unshaded) column on the right side is checked. Each of the 4 columns designates a CAM feature. If any one box in a column is checked, the feature is considered present. The CAM algorithm is considered positive if the following features are present: Feature 1) Acute onset or fluctuating course and Feature 2) Inattention and either Feature 3) Disorganized thinking or Feature 4) Altered level of consciousness.

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Garcia, MD PhD, Principal Investigator — Columbia University
Locations (1):
- NewYork-Presbyterian Allen Hospital/CUMC Milstein Hospital Building, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared in aggregate form. There is no plan to share individual participant data (IPD) with researchers not involved with the study design. Several posthoc analyses are being planned for retrospective analysis of the data obtained.